CLINICAL TRIAL: NCT06989619
Title: Leveraging Social Networks to Improve Sleep and Mindfulness Among Older Adults in Residential Housing Facilities
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Rebecca Robbins, Assistant Professor, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BrighamHopsital; R34AG089176 (NIH)
Record Dates: First submitted 2025-05-04; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Aging; Cognitive Impairment; Sleep
Keywords: Sleep health; Healthy lifestyle; Behavioral intervention
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sleep Health and Mindfulness Program for Older Adults (Experimental): This grant will develop and design an adapted version of an existing, effective Sleep Health Program, which will be coupled with mindfulness content, to meet the needs and unique barriers older adults in housing facilities face. The modules for the proposed Sleep Health and Mindfulness program will be designed in collaboration with the implementation partner, the City of Boston Age Strong Commission, whose talented leaders and staff have decades of experience designing programs for seniors on a variety of topics, including mindfulness.
  Interventions: Behavioral: Sleep health and mindfulness intervention

INTERVENTIONS:
Behavioral: Sleep health and mindfulness intervention — This educational, healthy lifestyle intervention will include several modules detailing sleep health and mindfulness strategies. In addition, opinion leaders will be identified in the population to help diffuse messages through each housing facility.

SUMMARY:
The aim of this study is to design a sleep and mindfulness intervention to improve sleep, quality of life, and cognitive function among older adults.

DETAILED DESCRIPTION:
The proposed R34 planning grant will the design and adapt a sleep, mindfulness, and sleep disorders education intervention entitled to cognitively unimpaired older adults residing in housing facilities. Novel, social network techniques will be used to identify opinion leaders who will assist with message dissemination. This grant will adapt content from an existing, evidence-based Sleep Health Program to the needs of older adults. In addition, the adapted Sleep Health Program will be coupled with Mindfulness content then disseminated in a small pilot study to ascertain feasibility and acceptability of the proposed novel social network approach for deploying the adapted Sleep Health and Mindfulness Program in a planned R01. The data collected in this R34 will include qualitative interview and usability interview data where cognitively unimpaired older adults will be recruited and asked to provide input to the messages and approach. Target outcomes will also be collected in the planned pilot, including survey responses to sleep, sleep disorders evaluation/care, quality of life, and cognition. Finally, FitBit data will also be captured for 2 weeks at several time points during the pilot study (baseline, 2-months, and 6-months).

ELIGIBILITY:
Inclusion Criteria:

* Older adults (age 55 years of age and above) residing in residential facilities.

Exclusion Criteria:

* Severe cognitive impairment according to the Montreal Cognitive Assessment (MoCA).

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Time it takes to recruit | Baseline, 2-months, and 6-months
  Time it takes to recruit participants into the study
Sessions attended | Baseline, 2-months, and 6-months
  Average number of sessions the participants attend.
Proportion of participants who complete the program | Baseline, 2-months, and 6-months
  Proportion of older adults who complete the program.

SECONDARY OUTCOMES:
The score of the Pittsburgh Sleep Quality Index (PSQI) | Baseline, 2-months, and 6-months
  The Pittsburgh Sleep Quality Index (PSQI) contains 19 self-rated questions which measures seven aspects of sleep: (1) subjective sleep quality, (2) sleep latency, (3) sleep duration, (4) habitual sleep efficiency, (5) sleep disturbances, (6) use of sleeping medication, and (7) daytime dysfunction. The 19 self-rated items are combined to form seven component scores, each of which has a range of 0-3 points (0 indicates no difficulty, while 3 indicates severe difficulty). The seven component scores are then summed to yield one global score, with a range of 0-21 points (0 indicating no difficulty, and 21 indicating severe difficulties in all the seven areas of sleep quality).
The Score of the Dementia Quality of Life (DEMQOL) | Baseline, 2-months, and 6-months
  The Dementia Quality of Life (DEMQOL) instrument is a 28-item self-reported measure related to health-related quality-of-life (HRQL) in patients with dementia. The DEMQOL takes cognition, negative emotion, positive emotion, social relationships, and loneliness into consideration.
The Score of the Montreal Cognitive Assessment (MoCA) | Baseline, 2-months, and 6-months
  The MoCA (Montreal Cognitive Assessment) test is scored out of 30 points, and a score of 26 or above is generally considered normal. A score of 26 or below may indicate some degree of cognitive impairment. The specific cutoff score for determining impairment is 26.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Robbins, PhD, Study Chair — PhD
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
All data collected in this R34 will be fully anonymous. Data and metadata will be made available through the NIH-funded National Sleep Research Resource (NSRR; www.SleepData.org). Data and metadata will be assigned a unique Digital Object Identifier (DOI) and a formal study citation by the repository (NSRR). All de-identified data will be shared by end of project period or time of publication, whichever is sooner, and will remain available indefinitely. We estimate data will be shared no later than year 2 of this R34 planning grant.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: All de-identified data will be shared by end of project period or time of publication, whichever is sooner, and will remain available indefinitely. We estimate data will be shared no later than year 2 of this R34 planning grant.
Access Criteria: Consistent with the Brigham and Women's Hospital data sharing guidelines